CLINICAL TRIAL: NCT04461665
Title: Effects of Vitamin D Supplementation on Immune Function in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shih Chien University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150301R
Record Dates: First submitted 2017-07-24; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D, immune, infants, breastfeeding
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: 4 months old or 6 months old breastfeeding infants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Enroll 6 months old breast feeding infant, who have not supplement vitamin D at pediatric clinic.
- VitD supplement (Experimental): Enroll 4 months old breast feeding infant, and provide 10 μg vitamin D daily for 2 months.
  Interventions: Other: vitamin D

INTERVENTIONS:
Other: vitamin D — vitamin D supplement 10 μg daily for 2 months
  Other Names: Baby Ddrops® Liquid Vitamin D3 Vitamin Supplement
  Arms: VitD supplement

SUMMARY:
Current study shows that vitamin D deficiency might affect human's immune function. Although breast milk is the best food of infants, however the vitamin D content in breast milk is low. Thus, breastfeeding infants are at high risk of vitamin D deficiency.Children's development and health are always the most important issues for parents. However, high prevalence of allergy in infants in Taiwan were not only with environmental factor which may also relate to their nutritional status. The aim of this study was to enroll breastfeeding infant at age of 4 month, and provide vitamin D supplement 10 μg daily until 6 month, to discuss the effects of vitamin D supplementation on immune function in infants.

DETAILED DESCRIPTION:
Study plan to enroll breastfeeding infant at age of 4 month, and provide vitamin D (vitD) supplement 10 μg daily until 6 month. we also enroll 6 month-old infant as control group.

All infants collected 5 ml artery blood and measured vitD nutritional status and immune function. Blood analysis contain complete blood count (CBC), differential count (DC), serum calcium, serum Parathyroid hormone (PTH), serum 25(OH)D3, serum total immunoglobulinE (IgE) and cell phagocytosis.

Peripheral blood mononuclear cell (PBMC) in blood was separated and cultured with complete medium contain 10% fetal bovine serum (CM10), or with different mitogens, include lipopolysaccharide (LPS), phorbol 12-myristate 13-acetate and ionomycin (PI) and house dust mite extract (HDM). PBMC are incubated at 37 ℃, 5% CO2 for 48 hours, and determined the expression of B cell with IgE receptor CD21 and CD23 and T regulatory cell with transcription factor Foxp3 by flow cytometry. All data were analyzed with SPSS 20.0. Infant sex and feeding type were analyzed by chi-square analysis. Difference between vitD supplement group and control group were analyzed by student's t test. Relationship between 25(OH)D3 and Calcium or PTH were analyzed by pearson correlation analysis. There was a significant difference when p-value was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding healthy infants

Exclusion Criteria:

* heart disease
* liver disease
* lung disease
* Intestinal disease

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Characteristic of infants-1 | Infants at 4 months old
  Gender in baseline
Characteristic of infants-2 | Infants at 4 months old
  Gestational week (week) in baseline
Characteristic of infants-3 | Infants at 4 months old
  Birth length (cm) in baseline
Characteristic of infants-4 | Infants at 4 months old
  Birth weight (kg) in baseline
Characteristic of infants-5 | Infants at 4 months old
  Birth head circumference (cm) in baseline
Characteristic of infants-6 | Infants at 4 months old
  Exposed to the sun (min/day) in baseline
Characteristic of infants-7 | Infants at 4 months old
  Exclusive breast-fed n (%) in baseline
Characteristic of infants-8 | Infants at 4 months old
  Mixed-fed n (%) in baseline
The anthropometric of infants from 4 months old to 6 months old-1 | Infants at 4 and 6 months old
  Length percentile (%) in both groups
The anthropometric of infants from 4 months old to 6 months old-2 | Infants at 4 and 6 months old
  Weight percentile (%) in both groups
Vitamin D nutritional status of infants-1 | Infants at 4 and 6 months old
  Ca (mg/dL) in both groups
Vitamin D nutritional status of infants-2 | Infants at 4 and 6 months old
  PTH (pg/mL) in both groups
Vitamin D nutritional status of infants-3 | Infants at 4 and 6 months old
  25(OH)D3 (ng/mL) in both groups

SECONDARY OUTCOMES:
Cell markers expression of B cells | Infants at 6 months old
  D21 and CD23 expression (%) in both groups
Cell markers expression of T cells | Infants at 6 months old
  Foxp3 expression (%) in both groups
Serum immunoglobulin E level of infants | Infants at 6 months old
  Concentration of IgE (ng/ml) in both groups
Cytokine levels in supernatant of lymphocyte by CM-10 induction-1 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-6 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by CM-10 induction-2 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-4 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by CM-10 induction-3 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-13 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by CM-10 induction-4 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-10 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by CM-10 induction-5 | Lymphocyte isolation from Infants at 6 months old
  Concentration of TGF-β (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by LPS induction-1 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-6 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by LPS induction-2 | Lymphocyte isolation from Infants at 6 months old
  Concentration of TNF-α (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by PI induction-1 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-4 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by PI induction-2 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-13 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by PI induction-3 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-10 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by PI induction-4 | Lymphocyte isolation from Infants at 6 months old
  Concentration of TGF-β (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by HDM induction-1 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IFN-γ (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by HDM induction-2 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-4 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by HDM induction-3 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-13 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by HDM induction-4 | Lymphocyte isolation from Infants at 6 months old
  Concentration of IL-10 (pg/ml) in both groups
Cytokine levels in supernatant of lymphocyte by HDM induction-5 | Lymphocyte isolation from Infants at 6 months old
  Concentration of TGF-β (pg/ml) in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Ming Chen, MD/PHD, Study Chair — Shih Chien University
Locations (1):
- Shih Chien University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasiliou JE, Lui S, Walker SA, Chohan V, Xystrakis E, Bush A, Hawrylowicz CM, Saglani S, Lloyd CM. Vitamin D deficiency induces Th2 skewing and eosinophilia in neonatal allergic airways disease. Allergy. 2014 Oct;69(10):1380-9. doi: 10.1111/all.12465. Epub 2014 Aug 4. PMID 24943330
- [Background] Chawes BL, Bonnelykke K, Jensen PF, Schoos AM, Heickendorff L, Bisgaard H. Cord blood 25(OH)-vitamin D deficiency and childhood asthma, allergy and eczema: the COPSAC2000 birth cohort study. PLoS One. 2014 Jun 12;9(6):e99856. doi: 10.1371/journal.pone.0099856. eCollection 2014. PMID 24925304
- [Background] Dawodu A, Davidson B, Woo JG, Peng YM, Ruiz-Palacios GM, de Lourdes Guerrero M, Morrow AL. Sun exposure and vitamin D supplementation in relation to vitamin D status of breastfeeding mothers and infants in the global exploration of human milk study. Nutrients. 2015 Feb 5;7(2):1081-93. doi: 10.3390/nu7021081. PMID 25665158
- [Result] Somashekar AR, Prithvi AB, Gowda MN. Vitamin d levels in children with bronchial asthma. J Clin Diagn Res. 2014 Oct;8(10):PC04-7. doi: 10.7860/JCDR/2014/10387.5055. Epub 2014 Oct 20. PMID 25478419